CLINICAL TRIAL: NCT01435083
Title: Desmopressin Melt Therapy in Patients With Nocturnal Polyuria: a Pharmacokinetic/Dynamic Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011/566
Record Dates: First submitted 2011-09-13; First posted 2011-09-15 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Nocturnal Polyuria
Keywords: Nocturia
MeSH Terms: conditions — Nocturia | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nocturnal polyuria patient with desmopressin MELT (Experimental)
  Interventions: Drug: Desmopressin

INTERVENTIONS:
Drug: Desmopressin — 120 µg, oral lyophilisate, sublingual use
  Other Names: Minirin Melt 120 µg, H01BA02

SUMMARY:
The objective of this study is to find out what the pharmacokinetic/dynamic (PK/PD) characteristics of desmopressin melt are in nocturia patients (compared to healthy volunteers and children). The main questions the investigators want to answer are:

* Are differences related to the pathophysiological factors involved in nocturia?
* Are there age/gender/size differences?
* Can the investigators identify patients who are likely to develop hyponatraemia?
* Can the investigators individualize treatment and reduce risk for hyponatraemia?

Day 1:

* Patient is being hospitalized in the morning
* General anamnesis and clinical examination
* Uroflow and residue measurements (3x)
* Sober blood sample, to determine plasma concentrations of Na+, Cl-, osmolality and creatinin

Day 1-2:

- In the evening at 20h:

* start (with empty bladder!) 24h miction-incontinence-residue registration: urine collections every 3 hours (every portion of urine within a period of 3 hours must be collected in the same collection device), with: registration of volumes and measurement urinary concentrations of Na+, Cl-, osmolality and creatinin
* Measurement of blood pressure during 24h

Day 2-3:

* In the evening at 19h (day 2): drink 15mL/kg water
* At 20h: take desmopressin melt 120µg + start:

  * 24h miction-incontinence-residue registration: registration of volumes and measurement urinary concentrations of Na+, Cl-, osmolality and creatinin (U1-U7)
  * Measurement of blood pressure during 24h
  * Collection of urine:U1 at 19h, U2 at 20h, together with intake of first desmopressin melt, U3 at 21h = 1h after desmopressin melt intake, U4 at 22h = 2 after desmopressin melt intake,U5 at 23h = 3h after desmopressin melt intake, U6 at 2h (day 3) = 6h after desmopressin melt intake, U7 at 8h = 12h after desmopressin melt intake
  * Blood samples for blood levels of desmopressin: 1h, 2h, 3h, 6h after desmopressin melt intake, 12h after desmopressin melt intake + plasma concentrations of Na+, Cl-, osmolality and creatinin (safety profile)
  * At 8h in the morning (day 3): drink 15mL/kg water + collection of urine per hour during 3h with measurement of urinary concentrations of Na+, Cl-, osmolality and creatinin: U8 at 9h, U9 at 10h, U10 at 11h
* Patient can go home on day 3, unless he is at high risk for side effects, high-risk patients are hospitalized for 7 days

ELIGIBILITY:
Inclusion Criteria:

* written informed consent prior to the performance of any study-related activity
* patients, men and woman, 18 years and older, with nocturnal polyuria, resulting in nocturia (2 voids or more at night) and/or nocturnal incontinence.

Exclusion Criteria:

* hypersensitivity/anaphylactic reaction on desmopressin or one of the other substances
* pregnancy
* genitourinary tract pathology (infection, tumor,...)
* urolithiasis
* suspicion or evidence of cardiac failure
* moderate to severe renal insufficiency (creatinin clearance < 50 ml/min)
* psychogenic or habitual polydipsia
* hyponatraemia or predisposition for hyponatraemia
* diabetes insipidus
* syndrome of inadequate ADH production

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic and dynamic evaluation of desmopressin melt for treatment of nocturnal polyuria in adults | hospitalisation of 3 days of which 15h specific for primary outcome measurements
  * blood analysis for plasma concentration of desmopressin: 1h, 2h, 3h, 6h and 12h after drug intake
  * urine analysis for urinary concentration of sodium, potassium, creatinin and osmolality:
    * after water load with 15ml/kg body weight (evening day 2): the moment of drug intake, 1h, 2h, 3h, 6h and 12h after drug intake
    * after water load with 15ml/kg body weight (morning day 3): 1h, 2h, 3h after water load

SECONDARY OUTCOMES:
24h miction-incontinence-residue registration: urine collections every 3 hours | 2x 24h: day 1 19h - day 2 19h ; day 2 20h - day 3 20h
  24h miction-incontinence-residu registration: urine collections every 3 hours (every portion of urine within a period of 3 hours must be collected in the same collection device), with:
  * Registration of volumes
  * Measurement urinary concentrations of Na+, Cl-, osmolality and creatinin
Measurement of blood pressure during 24h | 2x 24h: day 1 19h - day 2 19h ; day 2 20h - day 3 20h

CONTACTS AND LOCATIONS:
Overall Officials: Karel Everaert, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be